## Comparison of Kinesio Taping and Local Injection in Chronic Low Back Pain - NCT03895307

(08/01/2019)

## **Protocol:**

Approximately 84 volunteer patients will be included in the study, patients older than 18 years, under 75 years of age, with a minimum of 3 months of mechanical back pain, Visual Analog Scale score of at least 60 patients will be included. Who are older than 18 years of age, having mental problems, having peripheral problems affecting the central nervous system, having received physical therapy to the lumbar region in the last 3 months, having been applied to the lumbar region within the last 3 months, having a history of lumbar region surgery, having a history of patients with motor deficit in the extremity, needle phobia, lidocaine and / or kinesio tape allergy, patients with wound, infection, burn, allergic lesions in the application area will not be included.

Patients included in the study will be included in the first (first), second (second), third (third) or fourth (fourth) treatment group by random number generator method.

The first group will be given the hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16. days.

The second group will be given a hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16 days.

The third group hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16. days, kinesio tape will be applied to the determined areas.

the fourth group hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16. days sham tape application will be made in the regions determined.

Evaluations were made before treatment (T0), immediately after treatment (T1), 1 month (T2) and 3 months (T3) after treatment. Spinal mobility of the patients was measured in centimeters (cm) using the Schober test using a tape measure. VAS scored between 0-10 was used to evaluate the pain levels. Oswestry Disability Index (ODI) was used to evaluate the functional status of the patients. Short Form-36 (SF-36) questionnaire was used to evaluate the health-related quality of life of the patients.

## **Statistical Analysis:**

Statistical analyzes were performed using SPSS version 20 statistical software (IBM Corp., Armonk, NY). Average, standard deviation and frequency were used as descriptive statistical methods. Shapiro-Wilk and Kolmogorov-Smirnov tests were used to evaluate the distribution of numerical data. Since the data were not suitable for normal distribution, Mann Whitney U test was used to measure the difference between the group and Wilcoxon test was used to measure the temporal process. The differences between discrete variables were investigated by chi-square test. The results were evaluated in the 95% confidence interval and p <0.05 significance level.